CLINICAL TRIAL: NCT03652064
Title: A Phase 3 Study Comparing Daratumumab, VELCADE (Bortezomib), Lenalidomide, and Dexamethasone (D-VRd) With VELCADE, Lenalidomide, and Dexamethasone (VRd) in Subjects With Untreated Multiple Myeloma and for Whom Hematopoietic Stem Cell Transplant is Not Planned as Initial Therapy
Brief Title: A Study Comparing Daratumumab, VELCADE (Bortezomib), Lenalidomide, and Dexamethasone (D-VRd) With VELCADE, Lenalidomide, and Dexamethasone (VRd) in Participants With Untreated Multiple Myeloma and for Whom Hematopoietic Stem Cell Transplant is Not Planned as Initial Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108529; 54767414MMY3019 (Other: Janssen Research & Development, LLC); 2018-001545-13 (EudraCT Number); 2023-507312-13-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2018-08-17; First posted 2018-08-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bortezomib + Lenalidomide + Dexamethasone (VRd) and Rd (Active Comparator): Participants will receive bortezomib 1.3 milligram per square meter (mg/m^2) as subcutaneous (SC) injection twice weekly on Days 1, 4, 8, 11 for Cycles 1 through 8 (each cycle is of 21 days); lenalidomide 25 mg orally on Day 1 to Day 14 for Cycles 1 through 8 and on Days 1 to 21 for Cycle 9 (cycle of 28 days); dexamethasone 20 mg orally or intravenously on Days 1, 2, 4, 5, 8, 9, 11, 12 for Cycles 1 through 8 and 40 mg on Days 1,8, 15 and 22 during Cycle 9 and beyond (each cycle is of 28 days) followed by lenalidomide-dexamethasone (Rd) until disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Daratumumab + VRd (D-VRd) and DRd (Experimental): Participants will receive daratumumab 1800 mg as SC injection once every week for Cycles 1 to 2, then every 3 weeks for Cycles 3 through 8 and every 4 weeks for Cycle 9 and beyond; bortezomib 1.3 mg/m^2 as SC injection twice weekly on Days 1, 4, 8, 11 for Cycles 1 through 8 (each cycle is of 21 days); lenalidomide 25 mg orally on Day 1 to Day 14 for Cycles 1 through 8 and on Days 1 to 21 for Cycle 9; dexamethasone 20 mg orally or intravenously on Days 1, 2, 4, 5, 8, 9, 11, 12 for Cycles 1 through 8 and 40 mg on Days 1,8, 15 and 22 during Cycle 9 and beyond followed by daratumumab-lenalidomide-dexamethasone (DRd) until disease progression or unacceptable toxicity.
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab (1800 mg) will be administered by SC injection once every week for Cycles 1 to 2, then every 3 weeks for Cycles 3-8. For Cycle 9 and beyond, participants will receive daratumumab 1800 mg SC once every 4 weeks until documented disease progression or unacceptable toxicity.
  Other Names: JNJ-54767414; DARZALEX
  Arms: Daratumumab + VRd (D-VRd) and DRd
Drug: Bortezomib — Bortezomib 1.3 mg/m^2 will be administered by SC injection twice weekly on Days 1, 4, 8, and 11 of each 21-day cycle for Cycles 1-8.
  Other Names: Velcade
Drug: Lenalidomide — Lenalidomide will be self-administered at a dose of 25 mg orally on Day 1 to Day 14 for Cycles 1 through 8 and on Days 1 to 21 for Cycle 9 and beyond until disease progression or unacceptable toxicity whichever occurs first.
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone will be self-administered orally, 20 mg on Days 1, 2, 4, 5, 8, 9, 11, 12 of each 21-day cycle for Cycles 1-8. During Cycle 9 and beyond dexamethasone, will be self-administered orally at a total dose of 40 mg on Days 1, 8, 15, 22 of each 28-day cycle.

SUMMARY:
The purpose of this study to determine if the addition of daratumumab to bortezomib + lenalidomide + dexamethasone (VRd) will improve overall minimal residual disease (MRD) negativity rate compared with VRd alone.

DETAILED DESCRIPTION:
This study will evaluate participants with newly diagnosed multiple myeloma (MM) for whom hematopoietic stem cell transplant is not planned as initial therapy. The data available from other available studies suggests that addition of daratumumab with Velcade (bortezomib), lenalidomide, and dexamethasone [VRd] is anticipated to improve the response rates and the depth of response and may lead to improved long-term outcomes in newly diagnosed participants with MM. Daratumumab targets CD38, a protein expressed on the surface of MM cells and other hematopoietic cells. Bortezomib is a proteasome inhibitor, which plays a critical role in the pathogenesis of MM. Lenalidomide has cytotoxic effects on myeloma cells and is capable of inducing apoptosis, or programmed cell death and dexamethasone induces apoptosis in MM cells. The rationale for the study is to utilize the subcutaneous (SC) formulation of daratumumab instead of the intravenous (IV) formulation, which is expected to provide similar exposure and is expected to limit additional toxicity to participants, treated with this quadruplet regimen. The study will consist of 3 phases: Screening (up to 28 days before randomization), Treatment phase (from Cycle 1 [21 days] Day 1 and continues until disease progression) and Follow up (Postintervention). Efficacy evaluations will include measurements of tumor burden/residual disease, myeloma proteins, bone marrow examinations, skeletal surveys, extramedullary plasmacytomas, and serum calcium corrected for albumin. Participants will undergo procedures like electrocardiogram (ECG), chest x-rays or full dose chest CT scans, Pulmonary function test (PFT), spirometry etc. during the course of study. Participants will also be monitored closely for adverse events (AEs), laboratory abnormalities, and clinical response. The duration of the study will be approximately 6.5 years.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of multiple myeloma as documented per International Myeloma Working Group (IMWG) criteria Monoclonal plasma cells in the bone marrow greater than or equal to (>=)10 percentage (%) or presence of a biopsy proven plasmacytoma and documented multiple myeloma satisfying at least one of the calcium, renal, anemia, bone (CRAB) criteria or biomarkers of malignancy criteria. CRAB criteria: Hypercalcemia: serum calcium greater than (>) 0.25 millimoles per liter (mmol/L) (>1 milligram per deciliter [mg/dL]) higher than upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL); Renal insufficiency: creatinine clearance less than (<) 40 milliliter per minute (mL/min) or serum creatinine >177 micro millimoles per liter (umol/L) (>2 mg/dL); Anemia: hemoglobin >2 g/dL below the lower limit of normal or hemoglobin <10 g/dL; Bone lesions: one or more osteolytic lesions on skeletal radiography, computed tomography (CT), or positron emission tomography (PET)-CT.

Biomarkers of Malignancy: Clonal bone marrow plasma cell percentage >=60%; Involved: uninvolved serum free light chain (FLC) ratio >=100; >1 focal lesion on magnetic resonance imaging (MRI) studies

* Must have measurable disease, as assessed by central laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* A woman of childbearing potential must have 2 negative serum or urine pregnancy tests at Screening, first within 10 to 14 days prior to dosing and the second within 24 hours prior to dosing
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 3 months after receiving the last dose of any component of the treatment regimen

Exclusion Criteria:

* Frailty index of >=2 according to Myeloma Geriatric Assessment score
* Prior therapy for multiple myeloma other than a short course of corticosteroids (not to exceed 40 mg of dexamethasone, or equivalent per day, total of 160 mg dexamethasone or equivalent)
* Prior or concurrent invasive malignancy (other than multiple myeloma) within 5 years of date of randomization (exceptions are adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years)
* Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5
* Focal radiation therapy within 14 days of randomization with the exception of palliative radiotherapy for symptomatic pain management. Radiotherapy within 14 days prior to randomization on measurable extramedullary plasmacytoma is not permitted even in the setting of palliation for symptomatic management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Negative Minimal Residual Disease (MRD) Status | After randomization and prior to progressive disease (PD) or the start of subsequent anti-myeloma therapy approximately 2.5 years
  Percentage of participants who achieve MRD negative status by evaluation of bone marrow aspirates using next generation sequencing (NGS) at 10^-5 threshold will be assessed.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization to either disease progression or death whichever occurs first (approximately 6 years, or 9 years if the adaptive approach is decided at the interim)
  PFS is defined as the duration from date of randomization to either PD or death, whichever comes first. International Myeloma Working Group (IMWG) criteria for PD: Increase of 25 percentage (%) from lowest response value in any one of following: Serum M-component (absolute increase must be >= 0.5 gram per deciliter [g/dL],) Urine M-component (absolute increase must be >=200 mg/24 hours), participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase must be >10 milligrams per deciliter [mg/dL]), participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow PC% (absolute percentage must be >=10%), definite development of new bone lesions or soft tissue plasmacytomas or increase in size of bone lesions or tissue plasmacytomas and development of hypercalcemia (serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
MRD Negative Rate | 12,18 and 24 Months
  Percentage of participants who have achieved MRD negative status will be assessed and landmark timepoints (12, 18 and 24 months). MRD negativity will be evaluated as a potential surrogate for PFS and overall survival (OS) in multiple myeloma treatment.
Durable MRD Negative Rate | Throughout the study (approximately 6 year)
  Durable MRD negativity rate is defined as the number of participants who have achieved MRD negative status (at 10^-5) at 2 bone marrow aspirates examinations that are a minimum of 1 year apart, without any examination showing MRD positive status in between.
Overall Response Rate (ORR) | Up to the end of the study (approximately 6 years)
  ORR is defined as the percentage of participants who achieve partial response (PR) or better responses prior to subsequent anti-myeloma therapy in accordance with IMWG criteria, during or after the study treatment. IMWG criteria for PR: greater than or equal to (>=) 50 reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90 % or to less than (<) 200 mg/24 hours, If the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved free light chain (FLC) levels is required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow plasma cells (PCs) is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Very Good Partial Response (VGPR) or Better Rate | Approximately 6 years
  VGPR or better rate is defined as the percentage of participants achieving VGPR and complete response (CR) (including stringent complete response [sCR]) prior to subsequent anti-myeloma therapy in accordance with the IMWG criteria during or after the study treatment. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or greater than or equal to (>=) 90 % reduction in serum M-protein plus urine M-protein <100 milligram per 24 hours (mg/24 hours); CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% PCs in bone marrow. sCR: CR plus normal FLC ratio, and absence of clonal PCs by immunohistochemistry (IHC), immunofluorescence or 2- to 4 color flow cytometry.
Complete Response (CR) or Better Rate | Approximately 6 years
  CR or better rate is defined as the percentage of participants achieving CR or sCR prior to subsequent anti-myeloma therapy in accordance with the IMWG criteria during or after the study treatment.
PFS on the Next Line of Therapy | Time from randomization to progression on the next line of treatment or death, whichever comes first (up to approximately 6 years, or 9 years if the adaptive approach is decided at the interim)
  The PFS on the next line of therapy is defined as the time from randomization to progression on the next line of treatment or death, whichever comes first. Disease progression will be based on investigator judgment.
Overall Survival (OS) | From randomization until the participant's death from any cause (up to approximately 6 years, or 9 years if the adaptive approach is decided at the interim)
  OS is defined as the time from the date of randomization to the date of the participant's death due to any cause.
Time to Response | From randomization until PR or better until approximately 6 years
  Time to response is defined as the time between the randomization and the first efficacy evaluation at which the participant meets all criteria for PR or better.
Duration of Response (DOR) | From initial documentation of response to the date of PD until approximately 6 years
  DOR is calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of PD, as defined in the IMWG evaluation before the start of any subsequent anti-myeloma therapy.
Maximum Observed Serum Concentration (Cmax) of Daratumumab | Predose Cycle 1, Day 1 (C1D1), C3D1, C9D1, C12D1, and post dose C1D4, C3D4, Post-treatment Week 8 (Cycle 1 to 8 is of 21 days; Cycle 9 and onwards are of 28 days)
  The Cmax is the maximum observed serum concentration of daratumumab.
Minimum Observed Serum Concentration (Cmin) of Daratumumab | Predose, C1D1 (each cycle of 28 days), C3D1, C9D1, C12D1, and post dose C1D4, C3D4, Post-treatment Week 8 (Cycle 1 to 8 is of 21 days; Cycle 9 and onwards are of 28 days)
  The Cmin is the minimum observed serum concentration of daratumumab.
Number of Participants with Anit-daratumumab Antibodies | Predose, C1D1 (each cycle of 28 days), C9D1, C12D1, Post-treatment Week 8 (Cycle 1 to 8 is of 21 days; Cycle 9 and onwards are of 28 days)
  Number of participants with anti-daratumumab antibodies will be assessed.
Number of Participants with Anit-rHuPH20 Antibodies | Predose, C1D1 (each cycle of 28 days), C9D1, C12D1, Post-treatment Week 8 (Cycle 1 to 8 is of 21 days; Cycle 9 and onwards are of 28 days)
  Number of participants with anti-recombinant human hyaluronidase (rHuPH20) antibodies will be assessed.
Change from Baseline in Health-Related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 item (EORTC QLQ-C30) | Baseline, up to 6 years (end of study)
  The EORTC- QLQ-Core-30 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The recall period is 1 week ("past week") and responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A higher score represents greater HRQoL, better functioning, and more (worse) symptoms.
Change from Baseline in Health-Related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Multiple Myeloma 20-item (EORTC QLQ-MY20) | Baseline, up to 6 years (end of study)
  The EORTC QLQ-MY20 is a validated, self -administered instrument to assess QoL in persons with MM. This 20-item questionnaire measures the following domains: symptom scales, including disease symptoms (6 items) and symptoms related to side effects of treatment (10 items); function scale and future perspective (3 items); and body image (1 item).
Change from Baseline in HRQoL as Assessed by EuroQol Five Dimension Five Level Questionnaire (EQ-5D-5L) | Baseline, up to 6 years (end of study)
  The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The scores for the 5 separate questions are categorical and cannot be analyzed as cardinal numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (114):
- United States (19):
  - Innovative Clinical Research Inc, Cerritos, California
  - Baptist MD Anderson, Jacksonville, Florida
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Norton Healthcare, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Cancer And Hematology Centers of Western Michigan PC, Grand Rapids, Michigan
  - Saint Lukes Hospital Saint Lukes Cancer Specialists, Kansas City, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop, Mineola, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Good Samaritan Hospital Corvallis, Corvallis, Oregon
  - University Of Pittsburgh Medical Center UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Brazil (10):
  - Universidade Estadual De Campinas, Campinas
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Instituto Brasileiro de Controle do Cancer - Sao Camilo Oncologia, São Paulo
  - Hospital Santa Cruz, São Paulo
  - Clinica Medica Sao Germano S/S LTDA, São Paulo
- Canada (9):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - The Gordon & Leslie Diamond Health Care Center, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Brampton Civic Hospital, Brampton, Ontario
  - Victoria Hospital, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Quebec L Hotel Dieu de Quebec, Québec, Quebec
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Hemato-onkologicke oddeleni, Pilsen
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (8):
  - CHU Henri Mondor, Créteil
  - Centre Hospitalier Départmental La Roche sur Yon, La Roche-sur-Yon
  - Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Strasbourg Oncologie Libérale, Strasbourg
  - Institut Universitaire du cancer de Toulouse-Oncopole, Toulouse
- Germany (7):
  - phase 3 - Hämatoonkologischer Studienkreis am Klinikum Aschaffenburg, Aschaffenburg
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - St. Josef-Krankenhaus Hamm-Bockum-Hövel, Hamm
  - Institut für Versorgungsforschung, Koblenz
  - Universitatsmedizin Leipzig, Leipzig
  - Klinikum Großhadern der Ludwig-Maximilians-Universität, München
  - Universitaetsklinikum Tuebingen der Eberhard-Karls-Universitaet, Abteilung fuer Innere Medizin II,, Tübingen
- Israel (8):
  - Barzilai Medical Center, Ashkelon
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Med.Center - Hematology Institute, Haifa
  - Carmel Medical Center, Haifa
  - Meir Hospital, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky (Ichilov) Medical Center, Tel Aviv
- Japan (13):
  - Fukuoka University Hospital, Fukuoka
  - Ogaki Municipal Hospital, Gifu
  - Kanazawa University Hospital, Kanazawa
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - Matsuyama Red Cross Hospital, Matsuyama
  - Nagoya City University Hospital, Nagoya
  - National Hospital Organization Okayama Medical Center, Okayama
  - Japanese Red Cross Osaka Hospital, Osaka
  - National Hospital Organization Shibukawa Medical Center, Shibukawa
  - Japanese Red Cross Medical Center, Shibuya City
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - Albert Schweitzer ziekenhuis-lokatie Dordwijk, Dordrecht
  - Erasmus MC, Rotterdam
- Poland (10):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - NSSU Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Onkologii Ziemi Lubelskiej im sw Jana z Dukli, Lublin
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka, Słupsk
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Spain (6):
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hosp. Del Mar, Barcelona
  - Hosp. Univ. de Guadalajara, Guadalajara
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp. Mutua Terrassa, Terrassa
- Turkey (Türkiye) (7):
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara University School of Medicine Cebeci Hospital, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Ondokuz Mayis University, Samsun
- United Kingdom (9):
  - Monklands District General Hospital, Airdrie
  - Blackpool Victoria Hospital, Blackpool
  - University Hospital Wales, Cardiff
  - Colchester Hospital University NHS, Colchester
  - Leicester Royal Infirmary - Haematology, Leicester
  - Altnagelvin Hospital, Londonderry
  - The Royal Oldham Hospital, Oldham
  - Derriford Hospital, Plymouth
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Usmani SZ, Facon T, Hungria V, Bahlis NJ, Venner CP, Braunstein M, Pour L, Marti JM, Basu S, Cohen YC, Matsumoto M, Suzuki K, Hulin C, Grosicki S, Legiec W, Beksac M, Maiolino A, Takamatsu H, Perrot A, Turgut M, Ahmadi T, Liu W, Wang J, Chastain K, Vermeulen J, Krevvata M, Lopez-Masi L, Carey J, Rowe M, Carson R, Zweegman S. Daratumumab plus bortezomib, lenalidomide and dexamethasone for transplant-ineligible or transplant-deferred newly diagnosed multiple myeloma: the randomized phase 3 CEPHEUS trial. Nat Med. 2025 Apr;31(4):1195-1202. doi: 10.1038/s41591-024-03485-7. Epub 2025 Feb 5. PMID 39910273